CLINICAL TRIAL: NCT02938091
Title: Hepatic Lipase Variant -514 C/T in a High Fat vs. Low Fat Diet for Cardio-metabolic Outcomes: A Crossover Randomized Dietary Intervention Trial
Brief Title: Dietary Modulation of Hepatic Lipase (LIPC) -514 C/T Variant Associations With Lipids and Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Jose Ordovas, Director, Nutrition and Genomics Laboratory, Tufts University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Study 2480
Record Dates: First submitted 2016-10-16; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Dyslipidemia; Impaired Glucose Tolerance
Keywords: Hispanics; Single nucleotide polymorphism; Hepatic lipase
MeSH Terms: conditions — Dyslipidemias; Glucose Intolerance | interventions — Diet, High-Fat; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-fat diet (Experimental): The dietary intervention was designed as a typical Western diet (39% total fat, 14% saturated fat, 12% monounsaturated fat, 9.6% polyunsaturated fat, 42% carbohydrate, 8.8 grams fiber/1000 kcal)
  Interventions: Other: High-fat diet
- Low-fat diet (Experimental): The dietary intervention consisted of a Hispanic diet (20% total fat, 5.5% saturated fat, 9.6% monounsaturated fat, 3.7% polyunsaturated fat, 61% carbohydrate, 13.7 grams fiber/1000 kcal). The diet was comprised of typical foods and recipes resembling a traditional Caribbean Hispanic diet and differed from the Western diet in four primary ways: 1) more fruits and vegetables, 2) more beans (e.g. mixed dishes to reduce serving size of white rice while increasing legumes), 3) emphasis on reduced-fat dairy products (e.g., 1% fat milk), and 4) lower total fat and lower animal and hydrogenated fat.
  Interventions: Other: Low-fat diet

INTERVENTIONS:
Other: High-fat diet — Typical Western diet
  Arms: High-fat diet
Other: Low-fat diet — Traditional Caribbean Hispanic diet
  Arms: Low-fat diet

SUMMARY:
The investigators evaluated dietary modulation of LIPC rs1800588 (-514 C/T) for lipids and glucose using a randomized cross-over design comparing a high-fat Western diet and a low-fat traditional Hispanic diet in Caribbean Hispanics (n=42; 4 weeks/phase).

DETAILED DESCRIPTION:
The LIPC -514 C/T single nucleotide polymorphism (SNP) has been inconsistently associated with high density lipoprotein cholesterol (HDL-C) in population studies, supporting the possibility of its modulation by dietary factors. To investigate the interaction between the common LIPC -514(C/T) SNP and dietary fat, the investigators compared changes in lipids and glucose in response to two levels of dietary total fat (20% energy intake vs. 39% energy intake) in a crossover, randomized dietary intervention study enrolling Caribbean Hispanics. Individuals were screened for LIPC rs1800588 genotype prior to enrollment, and genotype-associated differences in response to diet were evaluated.

The study was designed to test the following hypotheses:

1. Carriers of the T allele consuming a low fat (LF) diet will have decreased hepatic lipase activity as compared with subjects with the CC genotype at the -514(C/T) polymorphism. Conversely, in individuals consuming a high fat (HF) diet, T carriers will exhibit an impaired ability to down regulate hepatic lipase activity.
2. Based on differences in hepatic lipase activity, the investigators hypothesized that a significant and clinically relevant proportion of the individual variability in fasting plasma HDL-C responses to changes in dietary fat intake would be due to variability at the LIPC locus. Specifically, CC subjects will respond to increases in total dietary fat consumption with significant increases in HDL-C concentration. Conversely, increased fat consumption in T carrying subjects will result in decreased HDL-C concentration.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Caribbean Hispanics

Exclusion Criteria:

* diabetes
* uncontrolled hypertension
* self-reported liver disease; severe kidney dysfunction; angina; endocrine disease; preexisting cardiovascular disease or gallbladder disease, or pancreatitis within the past 12 months
* use of lipid-lowering or hypoglycemic medications
* BMI >34 kg/m2
* alcohol consumption (>2 drinks/day)
* smoking within the past 6 months or illegal drug use
* pregnancy or breastfeeding
* weight gain or loss of more than 9 kg within the past 6 months
* extreme levels of physical or athletic activity, strict vegetarians/vegans
* egg, wheat, milk, fish, or nut allergies
* unwillingness to discontinue fish oil or flaxseed supplements or drinking alcohol during the study
* travel plans precluding availability for the two 4-week study phases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change in fasting high-density lipoprotein cholesterol | From date of randomization until completion of each 4 week dietary intervention

SECONDARY OUTCOMES:
change in fasting plasma triglycerides | From date of randomization until completion of the 4 week dietary intervention
change in fasting plasma glucose | From date of randomization until completion of the 4 week dietary intervention
oral glucose tolerance test | 2 hours post-oral glucose load
post-prandial lipemia 4 hours | 4 hours post-oral fat load
post-prandial lipemia 8 hours | 8 hours post-oral fat load

IPD SHARING:
Plan to Share IPD: No